CLINICAL TRIAL: NCT06525337
Title: Adherence of Health Coaching with Wearable Device
Brief Title: Adherence to Health Coaching with Wearable Devices: Enhancing Patient Engagement and Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coastal Carolina University (Other)
Collaborators: Apnimed (Industry); inHealth Medical Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024.182
Record Dates: First submitted 2024-07-09; First posted 2024-07-29 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; telehealth; AHI; Oxygen Saturation; ODI
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: All participants were randomized in a balanced fashion and stratified by sex and AHI number into either one of the two intervention groups STANDARDCARE group (STAND) compared to no sleep ring and health coaching CONTROL group (CON) group
Who Masked: Care Provider
Masking Description: Individuals will be randomized to the intervention or control at the baseline. SAS version 9.4 will be used to create the randomization list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STANDARDCARE (STAND) group (Experimental): Participants will download the Apnimed App for daily sleep ring data collection, using it nightly and syncing data each morning. They will receive weekly video health coaching sessions for 6 weeks, focusing on sleep, nutrition, and CPAP adherence. Surveys will be completed at baseline, 6 weeks, and 3 months.
  Interventions: Behavioral: STANDARDCARE (STAND) group
- CONTROL (CON) group (Experimental): Participants in this group will receive no device and no health coaching.
  Interventions: Other: CONTROL (CON) group

INTERVENTIONS:
Behavioral: STANDARDCARE (STAND) group — Will receive a device and health coaching
  Arms: STANDARDCARE (STAND) group
Other: CONTROL (CON) group — Will not use any devices or receive health coaching
  Arms: CONTROL (CON) group

SUMMARY:
The goal of this clinical trial is to learn how integrating health and wellness coaching (HWC) with Continuous Positive Airway Pressure (CPAP) therapy affects adherence to treatment and overall health outcomes in individuals with obstructive sleep apnea. The main questions it aims to answer are:

* Does HWC improve CPAP adherence compared to standard care, in terms of device usage metrics (hours per night and days per month)?
* How does combining HWC with weight management influence CPAP adherence and weight loss?
* What are the differences in treatment outcomes between individuals receiving standard care and those receiving HWC?

Researchers will compare two groups:

* Standard Care Group: Participants receiving standard CPAP therapy without additional health coaching.
* HWC Group: Participants receiving CPAP therapy combined with health and wellness coaching focused on weight management and sleep hygiene.

Participants will:

* Attend 2 in-office visits with a study physician (2 hours maximum)
* Have 6 virtual visits via video with a study health coach (3 hours maximum) if in the HWC group This study aims to provide valuable insights into enhancing treatment outcomes for individuals with sleep apnea by integrating health coaching with CPAP therapy.

DETAILED DESCRIPTION:
Purpose:

The purpose of this research study is to compare the effects of a wearable sleep ring combined with health coaching in the STANDARDCARE (STAND) group to a CONTROL (CON) group with no sleep ring and no health coaching. The investigators aim to see if this combination improves patient satisfaction and progress with using a CPAP machine.

Procedures:

If participants agree to participate, they will be asked to do the following:

Baseline Assessment:

Participants will attend a baseline assessment with their doctor that includes an overview and explanation of the study. They will conduct all standardized sleep tests as advised by their doctor. Upon meeting inclusion criteria, they will then be randomized to a STANDARDCARE (STAND) group or CONTROL (CON) group. During this time, body weight and height will be measured. Participants will then be asked to fill out several surveys that will involve questions related to overall health, quality of life, sleep adherence, and demographics (age, race).

STANDARDCARE GROUP (STAND):

If participants are randomized to this group, they will be asked to download one app. They will first be asked to download the Apnimed App, which will be used for collecting wearable sleep ring data daily. Participants will also be given step-by-step instructions on how to use the app. They will be asked to use the Apnimed sleep ring every night and sync data on the app in the morning. Following the initial baseline visit, participants will receive weekly individualized video health coaching sessions with a health coach through video conference using Zoom for 6 weeks. During these sessions, they will receive weekly educational online modules focusing on sleep, nutrition, and fitness centered on sleep science and adherence to the CPAP machine. Participants will be able to keep using the ring as much or as little as desired after the 6-week period. The research team will administer the final survey at 3 months following participants' first usage of the ring. Participants will fill out a survey at the beginning of the study, at 6 weeks, and 3 months after enrolling.

CONTROL GROUP (CON):

If participants are randomized to this group, they will not receive any wearable sleep ring or health coaching. They will have two visits with the study physician at baseline and at the end of the study. Participants will only be instructed to use the CPAP machine daily or undergo standard medical treatment as prescribed. They will be asked to fill out the surveys again at the end of 6 weeks and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Both genders
* All ethnicities
* Must reside in the state of TN
* Newly diagnosed with obstructive sleep apnea (OSA)
* Prescribed with moderate to severe OSA.7). AHI of > 15

Exclusion Criteria:

* Unable or unwilling to use wearable device,
* end stage renal failure
* heart failure or stroke
* Although not anticipated for this study population, women cannot be or suspect they may be pregnant.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-12-29 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Oxygen Desaturation Index (ODI) | Daily for 90 days
  The ODI is a measurement that helps diagnose and manage obstructive sleep apnea (OSA) by quantifying how often and how much a person's blood oxygen level drops during sleep.
Quality-of-life survey responses | Through Study Completion, an average of 3 months
  Quality-of-life survey responses assess an individual's overall well-being, encompassing physical, mental, and social health.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Williams Brice Building, Conway, South Carolina
  - Neurology Clinic, P.C., Cordova, Tennessee

IPD SHARING:
Plan to Share IPD: No